CLINICAL TRIAL: NCT01044849
Title: Clinical Test Report for Blood Pressure Meter CH-609
Status: Completed | Type: Observational
Sponsor: Citizen Systems Japan Co., Ltd. (Industry)
Responsible Party: Makoto Okamoto, Citizen Systems Japan Co., Ltd.
Other Study IDs: CH-609
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Blood Pressure
Keywords: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Blood pressure meter model CH-609 was to be assessed against the standard mercury sphygmomanometer according to the protocol of the ANSI/AAMI SP-10.

ELIGIBILITY:
Inclusion Criteria:

* 85 subjects with a wide range of blood pressure were selected.

Exclusion Criteria:

* Subjects could be taking antihypertensive medication, but excluded in atrial fibrillation or with any sustained arrhythmia.

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Measure the accuracy of blood pressure meter model CH-609 against the standard mercury sphygmomanometer according to the protocol of ANSI/AAMI SP-10. | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan